CLINICAL TRIAL: NCT01511744
Title: A Randomised, Controlled Phase IV Clinical Trial With an Inactivated Influenza Vaccine(Split Virion)
Brief Title: Phase IV Clinical Trial of an Inactivated Influenza Split Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Hualanbio-influenza IV-001; Hualanbio-phase IV-001 (Other Grant/Funding Number: Hualan Biological Engineering INC.)
Record Dates: First submitted 2012-01-18; First posted 2012-01-19 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-03

CONDITIONS: Human Influenza
Keywords: Respiratory Tract Infections; Orthomyxoviridae Infections
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inactivated influenza split vaccine (Experimental): Biological: Experimental: influenza split vaccine of 15 μg HA, one dose regime
  Interventions: Biological: Inactivated influenza split vaccine
- Blank control (No Intervention)

INTERVENTIONS:
Biological: Inactivated influenza split vaccine — 3000 participants (750 of above 60,750 of age 19-60, 750 of age 13-18 and 750 of age 3-12) to receive influenza split vaccine of 15 μg HA; one dose regime
  Other Names: Hualan Bio
  Arms: Inactivated influenza split vaccine

SUMMARY:
Influenza vaccine (split virion), Inactivated (15ug HA/subtype/0.5ml) of Hualan Biological Bacterin Co., Ltd (The subsidiary of Hualan Biological Engineering INC.) is applicable to the influenza immunity of age 3 and older population. Phase III clinical study was conducted in Jintan City, Jiangsu Province in May, 2006. Trial results showed that this vaccine had good safety and immunogenicity. Hualan Bio Influenza Vaccine obtained its production approval(China Drug Approval No.: S20083016) for marketing on April 3rd, 2008.

In order to monitor and evaluate the safety and protective effect against influenza administered on age 3 and older population, therefore we conduct the phase IV clinical trial of the licensed Influenza Vaccine (split virion), Inactivated (15ug HA/subtype/0.5ml).

DETAILED DESCRIPTION:
Select three sites to conduct this study in Henan, china. In the principle of informed consent and voluntary participation, adopt randomized and control design and include 6000 healthy subjects, among them, trial group 3000 persons, blank control group 3000 persons respectively and randomized dividing into 4 age groups.

The evaluation of safety: For all the vaccinated subjects, monitor general reaction and post-vaccination AEFI by mean of active soliciting and passive report. The evaluation of safety data mainly includes summary of clinical reaction endpoint, local and systemic adverse events of all subjects during the observation period and incidence rate of relevant ADR/AE.

The evaluation of immunogenicity: Respectively and randomly sample 600 persons from vaccination group and blank control group. Collect venous blood on the first day or 28 day of vaccination. Adopt international universal HI testing method(SRID) to carry out serology test.

The criteria for HI antibody test result:

* Take 1:10 serum as the lowest dilutability. For subjects whose HI antibody <1:10 before immunization, calculate as 1:5 and their post-vaccination HI antibody titer≥1:40 will be as the seroconversion. For subjects HI antibody ≥1:10 before the vaccination, take post-vaccination HI antibody titer increases 4 times as seroconversion;
* Take HI antibody titer≥1:40 as threshold of positive protection;
* Take statistics of subject number whose serum HI antibody titer reach protective level (HI antibody titer≥1:40). Calculate protection rate of vaccine and 95% CI;
* GMT titer and 95% CI. Evaluation of immune protective effect: Monitor Influenza Like Illness(ILI) to all subjects in monitoring place and conduct epidemiological survey to ILI. Collect nasopharyngeal swab and blood specimen during acute and recovery period for the laboratory test.

ILI refers to fever (body temperature≥38℃) with cough or pharyngalgia. Test influenza virus nucleic acid in nasopharyngeal swab. Isolate serum of blood specimen and carry out the test of serum antibody.

Evaluation indicator:

* Statistics of ILI incidence rate in immune population
* Statistics of incidence rate in monitoring place

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 3 and older, volunteers or their guardians are able to understand and sign the informed consent;
* Be able to abide by the requirement of clinical trial protocol to participate in follow up;
* Be willing to supply blood sample during clinical trial of vaccine and able to assist with filling out study data;
* Healthy male or female by inquiring illness history, physical examination and clinical judgment and who complies with vaccination of this product;
* Be able to comply with the requirement of clinical trial protocol;
* Have no history of vaccination and vaccination with other product in latest 1 week;
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Any history of severe illness, such as tumor, autoimmune disease, etc.;
* Subject that was allergic to any component of the vaccine (any history of vaccination allergy), especially eggs;
* History of neurological symptom or physical signs;
* Known or suspected (or high possibility of occurrence) damage of or abnormal immune function;
* Bleeding physique or prolonged bleeding;
* History of influenza infection or vaccination at least once within the past 6 months;
* History of administration of other vaccine or injection of immunoglobulin, or any research drug within the past 1 week;

  * Any acute disease that needs usage of antibiotics or antiviral therapy on the whole body within the past 7 days;
  * Fever (axillary temperature≥38℃) within the past 3 days;
* Participating in another clinical trial;
* History of Guillain-Barre Syndrome, severe birth defect or severe disease, allergy, eclampsia, epilepsy, encephalopathy or psychosis or family disease;
* Thrombopenia or other coagulopathy that may cause contraindication of intramuscular injection;
* Known or suspected other diseases at the same time, including respiratory system disease, acute infection or active period of chronic disease, HIV infection of infant or mother, cardiovascular disease, during of treatment of cancer and skin disease;
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety study | 28days
  Include ADR, adverse event, and severe adverse event.

SECONDARY OUTCOMES:
Observation of immune protective effect | 1year
  Observe immunogenicity and immune protective effect by means of active and passive monitoring. Period is one year.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Bianli, Master, Principal Investigator — Henan Province Center for Disease Prevention and Control
Locations (1):
- Henan Province Center for Disease Preventionand Control, Zhengzhou, Henan, China